CLINICAL TRIAL: NCT03471702
Title: A Secondary Study Evaluating Performance and Safety of Aqueduct's Smart External Drain (SED2)
Brief Title: A Secondary Study Evaluating Aqueduct's Smart External Drain (SED)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device Review performed by Sponsor
Sponsor: Aqueduct Critical Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASSESSED SED2
Record Dates: First submitted 2018-02-28; First posted 2018-03-21 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2018-03

CONDITIONS: Hydrocephalus; Hydrocephalus in Children; Tumor, Brain; Subarachnoid Hemorrhage
MeSH Terms: conditions — Hydrocephalus; Brain Neoplasms; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm Study (Experimental): All subjects enrolled on study will utilize Aqueduct's Smart External Drain (SED) from the time of external drain implementation until end of study upon discharge of SED or switch to standard of care external drain.
  Interventions: Device: Smart External Drain - SED

INTERVENTIONS:
Device: Smart External Drain - SED — Aqueduct's Smart External Drain (SED) is a gravity based system which utilizes a proprietary reference shroud which eliminates the need for manual adjustment of the system in the external management of CSF drainage.

SUMMARY:
Aqueduct's Smart External Drain (SED) will be compared to the current gold standard for temporary CSF management in a hospital setting.

* Evaluate the number of subjects requiring to be switched to a standard of care EVD
* Evaluate subject transport while on the SED
* Evaluate SED system control from initiation of SED through discharge of external drain system

DETAILED DESCRIPTION:
This clinical trial will evaluate Aqueduct's Smart External Drain (SED) upon implementation of ventriculostomy or lumbar drain placement for temporary CSF external management in a hospital setting. Subjects will remain on study from the time of SED application through discharge of the external drain or switch to standard of care extraventricular drain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject scheduled to have an external drain (includes extra-ventricular and lumbar drains) placed as part of routine management.
2. Age 0-80.
3. Able to obtain consent or legally authorized representative (LAR) consents for subject to be treated on study.

Exclusion Criteria:

1. Anticoagulant therapy (does not include DVT or PE prophylaxis).
2. Known bleeding diathesis.
3. Scalp infection.
4. In the opinion of the Investigator the subject is not a good study candidate.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The number of subjects which require switching to a standard of care external drain. | The study review and data collection period will begin at the time SED is connected to the ventriculostomy catheter until discharge of ventriculostomy catheter; when subject no longer requires an external drain, assessed up to 90 days.
  Evaluating the number of subjects which require switching to a standard of care external drain versus the number of subjects which remain on the SED until study completion or discharge of the external drain.

SECONDARY OUTCOMES:
Subject transport while on the SED system. | Subject transport review and data collection will begin when the patient is moved from their primary hospital bed location until they reach a new secondary location or are returned to the primary location. Assessed up to 90 days.
  Evaluating subject transport while on the SED system, specifically, the number of minutes a subject will require clamping of the drain while being transported.
Evaluating SED system control throughout duration of study. | The study review and data collection period will begin at the time SED is connected to the ventriculostomy catheter until discharge of ventriculostomy catheter; when subject no longer requires an external drain, assessed up to 90 days.
  SED system control will be evaluated from initiation of ICP management through discharge of the subject's external drain.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Browd, MD, PhD, Study Director — Aqueduct Critical Care, Inc.
Locations (3):
- United States (3):
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington School of Medicine, Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided